CLINICAL TRIAL: NCT03214809
Title: The Use of a Point-of-care Thoracic Ultrasound Protocol for Hospital Medical Emergency Teams
Acronym: METUS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow inclusion rate (partly due to Covid-19)
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NL61884.091.17
Record Dates: First submitted 2017-06-19; First posted 2017-07-12 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Dyspnea; Coma; Hypotension and Shock
Keywords: ultrasound; MET team; Concordance
MeSH Terms: conditions — Dyspnea; Coma; Hypotension; Shock

STUDY DESIGN:
Intervention Model Description: When the MET team arrives first assessment will be done according to the abcde algorithm. If immediate interventions are needed (intubation, CPR etc) this will be done first (and noted). After the abcde assessment an initial diagnosis is noted. In the even weeks the thoracic ultrasound protocol will be done, in the uneven weeks not. After the use of ultrasound various variables are noted.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Thoracic ultrasound protocol (Experimental): ABCDE algorithm with Thoracic ultrasound protocol
  Interventions: Diagnostic Test: ultrasound protocol
- No Thoracic ultrasound protocol (No Intervention): ABCDE algorithm without Thoracic ultrasound protocol

INTERVENTIONS:
Diagnostic Test: ultrasound protocol — after first assessment and treatment by the MET team, an Multi-organ ultrasound protocol will be run by the MET doctor
  Arms: Thoracic ultrasound protocol

SUMMARY:
Study to assess the possible effects of the use of a point-of-care thoracic ultrasound protocol for hospital medical emergency teams (MET)

DETAILED DESCRIPTION:
Rationale: Study to assess the possible effects of the use of a point-of-care thoracic ultrasound protocol for hospital medical emergency teams Objective: Concordance between MET diagnosis with and without the use of ultrasound with the chart review definitive diagnosis will be studied. Also other secondary endpoints will be evaluated.

Study design prospective, interventional study Study population: patients on the general wards in need treatment by the MET team Intervention (if applicable): When the MET team arrives first assessment will be done according to the abcde algorithm. If immediate interventions are needed (intubation, CPR etc) this will be done first (and noted). After the abcde assessment an initial diagnosis is noted. In the even weeks the thoracic ultrasound protocol will be done, in the uneven weeks not. After the use of ultrasound various variables are noted.

Main study parameters/endpoints:

Concordance between MET diagnosis with and without the use of ultrasound with the chart review definitive diagnosis will be studied.

Also other secondary endpoints will be evaluated.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

The use of ultrasound is without direct side effects in terms of radiation or other potential (non)physical disturbances.

There are no data on the effects of the use of ultrasound during MET calls. The MET team will first deliver acute care if necessary, the ultrasound protocol can be done within 10-15 minutes which is acceptable in terms of MET call care. The MET team physician can at any point decide to use the ultrasound if he/she thinks it is necessary.

In other circumstances (e.g. emergency department or intensive care units) point-of-care ultrasound is considered to be part of standard care.

The investigators will study the potential influence of ultrasound during MET calls in terms of accuracy of the initial diagnosis and whether ultrasound influences initial treatment, patients' disposition and so on, ultrasound is no treatment nor will be the use of ultrasound be decisive in the treatment of MET call patients in this study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients on the general wards in need of treatment by the MET team.

Exclusion Criteria:

* age (<18 years),
* pregnancy:

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2020-05-11 (Actual); Study Completion 2020-05-11 (Actual)

PRIMARY OUTCOMES:
Concordance between MET diagnosis with and without the use of ultrasound with the chart review definitive diagnosis will be studied | after 2-3 weeks
  final diagnosis will be determined by 2 independent experts on the basis of chart review and will be compared with the MET team diagnosis. There are 8 pre defined diagnosis categories. The difference in concordance between the MET diagnosis with and without the use of ultrasound with the definitive diagnosis will be tested with a chi-square or a Fisher Exact test in case of small expected frequencies.

SECONDARY OUTCOMES:
Possible difference in diagnostic certainty | direct after inclusion
  diagnostic certainty is measured on a scale 0-10. - Descriptive statistics will be presented as mean with standard deviation for normally distributed continuous data, median and inter-quartile range for skewed continuous variables. Differences between groups will be tested using the Students' T-test. In case of unevenly distributed variables, differences between groups will be tested using the Mann Whitney U Test.
Possible differences in initial treatment | direct after inclusion
  There are 11 pre-defined therapy categories. - Descriptive statistics will be presented as numbers and percentages for dichotomous and categorical variables. Differences between groups will be tested with a chi-square or a Fisher Exact test in case of small expected frequencies.
Possible differences in patients' disposition | direct after inclusion
  There are 4 pre-defined categories in patients' disposition. - Descriptive statistics will be presented as numbers and percentages for dichotomous and categorical variables. Differences between groups will be tested with a chi-square or a Fisher Exact test in case of small expected frequencies.
Whether the use of ultrasound was considered to be helpful | direct after inclusion
  The answer to this question is binary (yes or no). - Descriptive statistics will be presented as numbers and percentages for dichotomous and categorical variables. Differences between groups will be tested with a chi-square or a Fisher Exact test in case of small expected frequencies.
MET physicians characteristics | direct after inclusion
  there are 5 pre-defined categories in MET physician characteristics. - Descriptive statistics will be presented as numbers and percentages for dichotomous and categorical variables. Differences between groups will be tested with a chi-square or a Fisher Exact test in case of small expected frequencies.
Possible difference in the time needed to reach a diagnosis | direct after inclusion
  time in minutes. - Descriptive statistics will be presented as mean with standard deviation for normally distributed continuous data, median and inter-quartile range for skewed continuous variables. Differences between groups will be tested using the Students' T-test. In case of unevenly distributed variables, differences between groups will be tested using the Mann Whitney U Test.
Possible difference in the need for supervisor attendance | direct after inclusion
  the answer to this question is binary (yes or no). - Descriptive statistics will be presented as numbers and percentages for dichotomous and categorical variables. Differences between groups will be tested with a chi-square or a Fisher Exact test in case of small expected frequencies.
Number of times ultrasound was used in te "non-ultrasound weeks" | direct after inclusion
  answer to this question is a number. - Descriptive statistics will be presented as mean with standard deviation for normally distributed continuous data, median and inter-quartile range for skewed continuous variables. Differences between groups will be tested using the Students' T-test. In case of unevenly distributed variables, differences between groups will be tested using the Mann Whitney U Test

CONTACTS AND LOCATIONS:
Overall Officials: Michael Blans, MD, Principal Investigator — Rijnstate Hospital
Locations (1):
- Rijnstate Hospital, Arnhem, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blans MJ, Bousie E, van der Hoeven JG, Bosch FH. A point-of-care thoracic ultrasound protocol for hospital medical emergency teams (METUS) improves diagnostic accuracy. Ultrasound J. 2021 Jun 4;13(1):29. doi: 10.1186/s13089-021-00229-3. PMID 34089087